CLINICAL TRIAL: NCT03518398
Title: Effectiveness and Safety of Intense Pulsed Light in Patients With Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Yonrawee Piyacomn, M.D., FICO, Yonrawee Piyacomn, MD, FICO, Principal Investigator, Fellow of Cornea and Refractive Surgery Unit, Department of Ophthalmology, Faculty of Medicine, Chulalongkorn University, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yonrawee Piyacomn
Record Dates: First submitted 2018-04-16; First posted 2018-05-08 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Meibomian Gland Dysfunction (Disorder); Dry Eye Syndromes
Keywords: Intense pulsed light; Meibomian gland dysfunction; Dry eye; cytokines
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPL group (Experimental): IPL 9-13 J/cm2 according to Fitzpatrick's skin type on day 0, 15, 45
  Interventions: Device: Intense Pulsed Light; Combination Product: Standard treatment
- sham-IPL group (Sham Comparator): IPL 0 J/cm2 according to Fitzpatrick's skin type on day 0, 15, 45
  Interventions: Combination Product: Standard treatment

INTERVENTIONS:
Device: Intense Pulsed Light — E> Eye (E-SWIN, Paris, France) IPL machine
  Arms: IPL group
Combination Product: Standard treatment — warm compression, lid scrub and non-preservative ocular lubricants

SUMMARY:
Meibomian gland dysfunction (MGD) is one of the most common causes of dry eye diseases. Over the past decade, several treatment options in MGD have been extensively studied including warm compression, lid hygiene, ocular lubricants, forceful expression, LipiFlow thermal pulsation system, intraductal probing, debridement scaling and intense pulsed light (IPL). IPL is a broad spectrum, non-coherent and polychromatic light source with a wavelength spectrum of 500-1200 nm. It can be filtered to allow only a range of wavelengths to be emitted. Different wavelength makes different depth of tissue to absorb a specific light energy. Intense pulsed light (IPL) has been widely used in dermatology as a therapeutic tool for removal of hypertrichosis, benign cavernous hemangioma, benign venous malformations, telangiectasia, port-wine stain and pigmented lesions. Concurrent ocular surface improvements have been observed in patients undergone IPL treatment. Very few prospective clinical trials showed that subjective dry eye symptoms decreased and some of the dry eye signs also improved. Nonetheless, there is still inconsistency in the efficacy of IPL among these studies. Biomarkers, specifically cytokines, in dry eye diseases have been studied to some extent. Moreover, the change in ocular surface inflammatory cytokines in patients with MGD after IPL treatment is unclear.

The investigators proposed a prospective randomized double-masked sham-controlled clinical trial to investigate the efficacy and safety of intense pulse light in MGD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and sign an informed consent form
2. 18-80 years of age
3. Fitzpatrick skin type 1-5
4. Able and willing to comply with the treatment /follow-up schedule and requirements
5. Presence of meibomian gland on each lower eyelid's meibography
6. Current diagnosis of stage1-4 of MGD in both eyes, according to the International Workshop on Meibomian Gland Dysfunction: Report of the Subcommittee on Management and Treatment of Meibomian Gland Dysfunction

Exclusion Criteria:

1. Contact lens wearer within the past 1 month and throughout the study
2. Recent ocular surgery or eyelid surgery within the past 6 months
3. Neuro-paralysis in the planned treatment area within the past 6 months
4. Current use of punctual plugs
5. Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area
6. Uncontrolled infections or uncontrolled immunosuppressive diseases
7. Subjects who have undergone refractive surgery within the past 6 months
8. Diseases in the planned treatment area that could be stimulated by light at 560 nm to 1200 nm (e.g.,Herpes simplex 1 and 2, Systemic Lupus Erythematosus, porphyria)
9. Use of photosensitive medications and/or herbs that may cause sensitivity to 560-1200 nm light exposure, such as isotretinoin, tetracycline, or St. John's Wort
10. Pregnancy and lactation
11. Radiation therapy to the head or neck within the past year, or planned radiation therapy throughout study period
12. Treatment with chemotherapeutic agent within the past 8 weeks, or planned chemotherapy throughout study period
13. Any condition revealed during the eligibility screening process whereby the physician deems the subject inappropriate for this study
14. Declared legally blind in one eye
15. IPL treatment within the past 12 months
16. Lipiflow treatment, or any equivalent treatments, within the past 12 months
17. Any anti-glaucomatous eye drop uses within the past 3 months and throughout the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Change in fluorescein tear break-up time at month 6 using fluorescein technique | day 0, 15, 45, month 3, month 6
  time elapsed from the last complete eyelid blink until appearance of the first dry spot on the cornea

SECONDARY OUTCOMES:
Change in dry eye symptoms using Ocular Surface Disease Index (OSDI), a questionnaire, at month 6 | day 0, 15, 45, month 3, month 6
  a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning.
Change in lipid layer thickness at month 6 using LipiView interferometer (TearScience inc., Morrisville,NC) | day 0, 15, 45, month 3, month 6
  quantitative values of the tear-film lipid layer depth or thickness by imaging the surface contour of the tear film, lipid layer thickness measurement
Change in Meibomian gland's anatomy by Meiboscore using Meibography at month 6 using Keratograph 5M (OCULUS, Wetzlar, Germany) | day 0, 15, 45, month 3, month 6
  directly visualising the morphology of meibomian glands in vivo
Change in ocular surface staining at month 6 using fluorescein staining technique | day 0, 15, 45, month 3, month 6
  fluorescein dye which is a mildly invasive stain that marks the tear film and defects in the corneal and conjunctival epithelium. The investigators use National Eye Institute (NEI) grading for ocular surface staining score in this study
Change in Meibomian gland expressibility at month 6 after applying the force onto the eyelids using meibomian gland evaluator | day 0, 15, 45, month 3, month 6
  number of glands expressible after applying force onto the eyelids
Change in Meibum quality at month 6 after applying the force onto the eyelids using meibomian gland evaluator | day 0, 15, 45, month 3, month 6
  quality of the meibum content after applying the force onto the eyelids
Change in tear osmolarity at month 6 using TearLab Osmolarity System (San Diego, CA) | day 0, 45, month 3, month 6
  concentration of the tear : The investigators use TearLab Osmolarity System (San Diego, CA)
Change in tear production test (Schirmer's test) at month 3 using calibrated strips of a non-toxic filter paper | day 0, month 3
  is used determine whether the lacrimal glands produce enough tears to keep the eyes adequately moist
Change in tear cytokines Interleukins-1 receptor antagonist (IL-1Ra) at month 3 using Bio-Plex® 200 system (Bio-Rad, Hercules, CA) | day 0, month 3
  one of the tear inflammatory cytokines
Change in tear cytokines Interleukins-6 at month 3 using Bio-Plex® 200 system (Bio-Rad, Hercules, CA) | day 0, month 3
  one of the tear inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Yonrawee Piyacomn, MD, Principal Investigator — Department of Ophthalmology, Faculty of Medicine, Chulalongkorn University
Locations (1):
- Yonrawee Piyacomn, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No